CLINICAL TRIAL: NCT00428207
Title: Glycemic Stability of Insulin Aspart Versus Insulin Lispro in Insulin Pump Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Treatment differences not detected with 7 point fingerstick monitoring
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-18
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes, insulin pump therapy, glycemic stability
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Aspart Versus Insulin Lispro (Active Comparator): Insulin aspart will be used for diabetes management, and will be delivered continuously, subcutaneously using a pump for a four week period. Insulin aspart doses will be adjusted by the principal investigator as needed to maintain glycemic control. Insulin dose adjustments will vary from patient to patient based on the carbohydrate consumption, level of physical activity, and fingerstick monitoring results SMBG (7 times per day). SMBG results collected during this four week period will be compared to the SMBG results collected while participant uses alternative treatment (insulin Lispro).
  Interventions: Drug: Insulin Aspart versus Insulin Lispro
- Insulin Lispro Versus Insulin Aspart (Active Comparator): Insulin lispro will be used for diabetes management, and will be delivered continuously, subcutaneously using a pump for a four week period. Dose will be adjusted as needed to maintain glycemic control. Insulin dose adjustments will vary from patient to patient based on the carbohydrate consumption, level of physical activity, and fingerstick monitoring results SMBG (7 times per day). SMBG results collected during this four week period will be compared to the SMBG results collected while participant uses alternative treatment (insulin Aspart).
  Interventions: Drug: Insulin Lispro versus Insulin Aspart

INTERVENTIONS:
Drug: Insulin Aspart versus Insulin Lispro — Subjects will be randomly assigned to insulin aspart versus insulin lispro via random number generation. Half of the patients will begin with insulin aspart, and then will be crossed over to insulin lispro. The insulin sequence will be reversed for the other half of the patients.
  Other Names: NovoLog; NovoRapid; Humalog
  Arms: Insulin Aspart Versus Insulin Lispro
Drug: Insulin Lispro versus Insulin Aspart — Subjects will be randomly assigned to insulin lispro versus insulin aspart via random number generation. Half of the patients will begin with insulin lispro, and then will be crossed over to insulin aspart. The insulin sequence will be reversed for the other half of the patients.
  Other Names: Humalog; NovoRapid; Novolog
  Arms: Insulin Lispro Versus Insulin Aspart

SUMMARY:
The purpose of this study is to determine:

1. whether there is a difference between insulin aspart and insulin lispro in continuous insulin pump therapy
2. whether duration of the insulin infusion set placement effect blood sugar control if the infusion set is in place for longer then 72-96 hours

DETAILED DESCRIPTION:
Insulin instability in pump infusion systems can result in unexplained hyperglycemia in patients on continuous subcutaneous insulin infusion (CSII) therapy. We have noted that some pump patients develop glycemic instability with use of insulin lispro, and that this resolves with change to insulin aspart. Several patients using lispro have reported noting a whitish precipitate in the infusion set, and in two cases we have examined the catheters and confirmed biochemically that this precipitate was insulin. Furthermore, in vitro studies indicate that insulin aspart is more resistant to isoelectric precipitation than insulin lispro. Although it has been rare for patients to notice a visible precipitate in the pump catheter, there is a subset of patients using lispro who have noted that their blood glucose levels will tend to rise 2 or more days after the insertion of a new pump infusion system. These findings mirror bench studies showing that the relative stability differences between aspart and lispro in pump infusion systems becomes more apparent over time.

The endpoints examined in previous randomized clinical trials comparing aspart and lispro were not directed specifically at assessing the effect of insulin type on glycemic stability. In these previous studies, pump infusion systems were changed every 48 hours whereas most pump patients routinely replace their infusion catheters only every 72-96 hours; this discrepancy may account for the failure of these trials to demonstrate the difference in the stability of insulin aspart and lispro that has been noted in clinical practice.

This investigator-initiated clinical trial is intended to assess the safety and efficacy of CSII with insulin aspart compared to insulin lispro with use of pump infusion catheters for up to 96 hours.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes treated with CSII at least 3 months.
* Males and females, > 18 years but < 75 years old.
* Hemoglobin A1c ≤ 8.0 % at measurement taken at week 0 (screening visit).
* Duration of diabetes ≥ 12 months.
* Willingness to perform self-blood glucose monitoring several times/day.

Exclusion Criteria:

* Previous insulin precipitation in pump infusion catheters.
* Daily insulin requirements > 25% of pump reservoir capacity. (This would preclude the subject from using the pump infusion system for more than 3 days).
* Use of an insulin pump that does not have a downloadable record of basal and bolus doses.
* Known or suspected allergy to trial products.
* Pregnancy, breast-feeding, intention to become pregnant or inadequate contraception measures.
* Known or suspected alcohol or drug abuse.
* Impaired renal function with creatinine ≥ 1.7 mg/dl.
* Pronounced catheter site scarring.
* Chronic use of drugs that may influence glycemic control (e.g. steroids).
* Any other significant concomitant disease that would interfere with participation in and completion of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Wolpert, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Around November 2006, patients were recruited through physician recommendations and also patient lists from clinic. Patients were sent letters asking them to be in the study. Study visits took place in the clinic.
Pre-assignment Details: This was a crossover study, so patients all began in one arm and were then switched to the other arm.
Groups:
- Insulin Lispro: Subjects will be randomly assigned to one of the two insulins (insulin Lispro) by the statistician working in the study via random number generation.
  First Intervention- four weeks using insulin Aspart in the pump. Subjects will use their current basal rates, insulin to carb ratios and correction factors to dose insulin.
  After the four weeks of the first intervention have been completed subjects will be switched to insulin lispro, for the second intervention period.
  The sequence of interventions may be reversed due to random assignment of treatment.
- Insulin Aspart: Subjects will be randomly assigned to one of the two insulins (insulin Aspart) by the statistician working in the study via random number generation.
  First Intervention- four weeks using insulin Aspart in the pump. Subjects will use their current basal rates, insulin to carb ratios and correction factors to dose insulin.
  After the four weeks of the first intervention have been completed subjects will be switched to insulin lispro, for the second intervention period.
  The sequence of interventions may be reversed due to random assignment of treatment.
Period: Overall Study
Arm/Group | Insulin Lispro | Insulin Aspart
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All study participants received both interventions.
Groups:
- Insulin Aspart Versus Insulin Lispro: insulin Aspart versus insulin Lispro : Subjects will be randomly assigned to one of the two insulins by the statistician working in the study via random number generation. Half of the patients will begin with insulin aspart, and then will be crossed over to insulin lispro. The insulin sequence will be reversed for the other half of the patients.
  Period 1: four weeks using insulin aspart in the pump, followed by Period 2: four weeks using insulin lispro in the pump, or vice versa depending on randomization.
  insulin pump :
Arm/Group | Insulin Aspart Versus Insulin Lispro
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.25 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Stability
Description: Glycemic stability will be assessed by MAGE (Mean Amplitude of Glycemic Excursion)(5), M value of Schlichtkrull, standard deviation & coefficient of variation using 7 point finger stick blood glucose measurements performed 48-96 hours after insertion of the pump infusion catheter. Data collected 48 to 72 hours post-catheter insertion will be analyzed separately from the data collected 72 to 96 hours post-catheter insertion. The mean of the measurements taken throughout the study will be used for calculation of the primary endpoint.
Time Frame: 48 to 96 hours
Population: Data collection was "incomplete/insufficient" and therefore endpoint could not could not be evaluated
Arm/Group | Insulin Aspart Versus Insulin Lispro | Insulin Lispro Versus Insulin Aspart
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Frequency of Catheter Change
Description: Recorded by the subjects who will use a checklist to document the reason for the catheter change (routine, insufficient insulin in infusion system, unexplained hyperglycemia, catheter site irritation, suspected occlusion/kinking of catheter, loosening of catheter.
Time Frame: 48 to 96 hours
Population: Data collection was incomplete/insufficient and therefore end points could not be evaluated for this assessment.
Arm/Group | Insulin Aspart Versus Insulin Lispro
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 Week study treatment period
Description: Adverse Events will be 'self-reported' by study participants at each study visit in addition to potential AEs observed by the investigator on the study participant's study diary (logbook).
Groups:
- Insulin Aspart Versus Insulin Lispro: insulin Aspart versus insulin Lispro : Subjects will be randomly assigned to one of the two insulins by the statistician working in the study via random number generation. Half of the patients will begin with insulin aspart, and then will be crossed over to insulin lispro. The insulin sequence will be reversed for the other half of the patients.
  Period 1: four weeks using insulin aspart in the pump, followed by Period 2: four weeks using insulin lispro in the pump, or vice versa depending on randomization.
Arm/Group | Insulin Aspart Versus Insulin Lispro
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The 7 point fingerstick blood glucose profile was not sensitive enough to detect differences in the treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No